CLINICAL TRIAL: NCT01349699
Title: Effects of Iron Loading and Iron Chelation Therapy on Innate Immunity During Human Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Peter Pickkers, MD. PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2009/189
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Systemic Inflammatory Process; Anemia
Keywords: endotoxemia; inflammation; iron; iron chelation; cytokines
MeSH Terms: conditions — Anemia; Endotoxemia; Inflammation | interventions — Ferric Oxide, Saccharated; Deferasirox; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Iron loading (Active Comparator): Subjects will receive 1.25 mg/kg iron sucrose intravenously 1 hour before endoxin administration 2ng/kg.
  Interventions: Drug: iron sucrose; Drug: endotoxin
- Iron chelation (Active Comparator): Subjects will receive 30mg/kg deferasirox orally 2 hours before endotoxin administration 2ng/kg.
  Interventions: Drug: Deferasirox; Drug: endotoxin
- Placebo (Placebo Comparator): Subjects will receive placebo instead of iron chelation or iron loading before endotoxin administration
  Interventions: Drug: endotoxin; Drug: Placebo

INTERVENTIONS:
Drug: iron sucrose — 1.25 mg/kg iron sucrose is administered intravenously 1 hr before endotoxin administration
  Other Names: Venofer
  Arms: Iron loading
Drug: Deferasirox — 30 mg/kg deferasirox is administered orally 2 hrs before endotoxin administration.
  Other Names: Exjade
  Arms: Iron chelation
Drug: endotoxin — at t=0 2ng/kg purified E.Coli endotoxin is administered intravenously
  Other Names: LPS
Drug: Placebo — At t=-2 hrs starch is dissolved in water to serve as a placebo for exjade. It is prepared and administered orally by a research nurse that is unblinded to the protocol.
  At t=-1 hrs 0.9% NaCl is administered intravenously serving as a placebo for iron sucrose. The infused volume is identical, and the syringes en tubes are blinded by aluminum foil. The administration is carried out by a research nurse that is unblinded to the protocol.
  Arms: Placebo

SUMMARY:
Iron affects immunity. However, the exact effect of iron on the innate immune response is not known. Animal data suggest that iron administration induced oxidative stress which enhances the innate immune response, whereas iron chelation has the opposite effect. The investigators tested the hypothesis that administration of iron sucrose 1.25 mg/kg augments the innate immune response, and iron chelation by deferasirox 30 mg/kg attenuates the innate immune response during human experimental endotoxemia.

DETAILED DESCRIPTION:
Systemic inflammation is accompanied by profound changes in iron distribution, mainly under the influence of hepcidin, leading to sequestration of iron in macrophages of the reticuloendothelial system, and ultimately anemia of inflammation. This redistribution of iron may represent an effective defense mechanism against a variety of pathogens, that need iron for replication and growth. The fact that iron withholding strategy is such a highly conserved part of the innate immune response illustrates that iron homeostasis and immunity are closely related. Concordantly, several studies in animal models have revealed immune modulatory effects of both iron and iron chelation: Iron sucrose has been shown to potentiate the inflammatory response and associated mortality, while iron chelation appears to attenuate inflammation and improve outcome in murine models of inflammation and sepsis. The immune modulatory effects of iron supplements and chelators are mainly attributed to their ability to potentiate or reduce the formation of reactive oxygen species (ROS). A subfraction of non-transferrin bound catalytically active iron, labile plasma iron, is thought to be responsible as this free iron is able to easily donate or accept electrons, thereby fueling redox reactions. Oxidative stress is associated with propagation of the immune response, endothelial dysfunction, and contributes to the organ damage that occurs during systemic inflammation. In accordance, anti-oxidants exert anti-inflammatory effects. As such, iron chelation has been suggested to be a valuable adjuvant therapy during infection for two distinct reasons: inhibition of bacterial growth and protection of organs against inflammation induced oxidative stress.

Effects of iron status on the immune response has up till now mainly been investigated in in vitro and in animal models, often using supra-therapeutic dosages of iron donors or iron chelators. Data on the effect of iron loading and iron chelation during systemic inflammation in humans are lacking. The objectives of the present study were to investigate the acute effect of therapeutic dosages of iron loading and iron chelation therapy on iron homeostasis, oxidative stress, the innate immune response, and subclinical organ injury during systemic inflammation induced by experimental endotoxemia in humans in vivo.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* between 18 and 35 years of age

Exclusion Criteria:

* smoking
* use of prescription drugs
* febrile illness < 2 weeks before the study date
* abnormalities found at screening
* participation in another trial in the preceding 6 months
* iron disorders in the family

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
TNF-alfa | Level of TNF-alfa 90 minutes after endotoxin administration
  Level of TNF-alfa 90 minutes after endotoxin administration

SECONDARY OUTCOMES:
Cytokines | 24 hrs after the administration of endotoxin
  Levels of TNF-alfa, IL-6, IL-10 IL-1RA, ICAM and VCAM.
Oxidative stress | 24 hrs after the administration of iron / iron chelator / placebo
  Several parameters of oxidative stress are measured:
  TBARS,carbonyls,oxidative radical production of neutrophils, ferric reducing ability of plasma.
Hemodynamic response | 24 hours after the administration of endotoxin
  Hemodynamic sequelae of endotoxin administration are monitored (heart rate, blood pressure) and the response of fore arm vessels to the infusion of vasoactive medication (norepinephrine, acetycholine, and nitroglycerine) is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center